CLINICAL TRIAL: NCT04077827
Title: TIVA Versus Volatile Anesthetics Admnistration on Stress and Pain Levels During Autologous Fat Transfer in Breast Reconstruction, in a Day Care Center
Brief Title: TIVA Admnistration and Autologous Fat Transfer in Breast Reconstruction
Acronym: TIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Saint Savvas Anticancer Hospital (Other)
Responsible Party: Principal Investigator, Maria Kapritsou, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2834
Record Dates: First submitted 2019-08-23; First posted 2019-09-04 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Admnistration Fat Transfer; Autologous Fat Transfer; Breast Reconstruction; TIVA; volatile anesthesia; stress levels; pain levels
MeSH Terms: conditions — Breast Neoplasms | interventions — Propofol; Remifentanil; Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia (Experimental): The patients will recieve intravenous anesthesia (propofol-remifentanyl)
  Recommended dosage:
  Propofol: Induction dosage 1,5-2,5 mg/kg Remifentanyl: Induction dosage 0,5-1μg/min The preservation dosage will depend from patients' body weight, body height and BMI
  Interventions: Drug: Propofol
- volatile anesthesia (Experimental): The patients will recieve volatile anesthesia (desflurane-remifentanyl)
  Recommended dosage:
  Desflurane dosage 6-7 MAC Remifentanyl: Induction dosage 0,5-1μg/min The preservation dosage will depend from patients' body weight, body height and BMI
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Patients will be divided into 2 groups. The TIVA group (N = 23) will be administrated intravenous anesthesia (propofol-remifentanil), while to the DES group (N = 23) volatile anesthetics (desflurane-remifentanil)
  Other Names: remifentanyl; desflurane

SUMMARY:
The aim of the present study is to investigate the effect of intravenous anesthetics versus the administration of volatile anesthetics on stress and pain levels during autologous fat transfer for breast reconstruction in a Day Care Center.

DETAILED DESCRIPTION:
The sample of the study will be patients who will have Autologous Fat Transfer for Breast Reconstruction.

Patients will be divided into 2 groups. The TIVA group (N = 23) will be administrated intravenous anesthesia (propofol-remifentanil), while the DES group (N = 23) volatile anesthetics (desflurane-remifentanil).

Specifically, the TIVA group will include patients over 50 years of age with high risk of nausea / vomiting and postoperative delirium, as well as suspicion of malignant hyperthermia. Patients with cardiac and respiratory problems will be included in the DES group.

The following data will be collected in the Data Sheet: Patient Demographics (Gender, Age), Body Mass Index (Body Height- Body Weight). Simultaneously, the pain levels will be evaluated by VAS Optical Analogue Scale of VAS 0-10 in PACU, preoperatively and postoperatively, and perioperative pain levels will be assessed with CPOT scale (values 0-8).

Stress levels will be evaluated with 3 NAS questions: a. How sad do you feel right now? b. How anxious do you feel right now? and c. How optimistic do you feel right now?. The 3 NAS questions will also be given preoperatively and postoperatively to the ward. The sedation levels will be assessed by RASS scale (values +4 to -5) and the Bispectral Index (BIS). The level of patient's awareness will be assessed by GCS Scale (3 (indicating deep unconsciousness) and either 14 (original scale) or 15 (more widely used modified or revised scale)).

The presence or absence of nausea / vomiting and the appearance of immediate postoperative complications will be examined. Finally, post-operative stress will be examined with stress biomarkers, salivary ACTH hormone and salivary cortisol hormone.

ELIGIBILITY:
Inclusion criteria:

TIVA group

* patients with American Society of Anesthesiologists (ASA) PHYSICALSTATUS CLASSIFICATION SYSTEM I-III
* age >50 years
* high risk of nausea / vomiting
* high risk of postoperative delirium
* suspicion of malignant hyperthermia.

Volatile anesthesia

* patients with American Society of Anesthesiologists (ASA) PHYSICALSTATUS CLASSIFICATION SYSTEM I-III
* 20-70 years
* Patients with cardiac problems
* Patients with respiratory problems

Exclusion Criteria

•In both groups, the exclusion criteria are the opposite of the inclusion criteria

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Εvaluating stress levels | 1 day during hospitalization
  Analyzing Cortisol and Adrenocorticotropic hormones levels in salivary samples.
  Analyzing Cortisol and Adrenocorticotropic hormones levels in salivary samples in patients after breast recostruction in a day care center.
  These measures will occured in three phases a. preoperatively, b. perioperatively c. in the PACU phase.

SECONDARY OUTCOMES:
Evaluating pain levels between the 2 protocols with scales perioperatively | 1 day during hospitalization
  Evaluating perioperative pain levels between the two protocols with scale such as Critical Care Pain Observational Tool (CPOT scale, range 0-8(with a score of 0 = None and 8 = severe pain) )
Evaluating stress levels between the 2 protocols with scales | 1 day during hospitalization
  Evaluating perioperative stress levels between the two protocols with scale, such as the self-experienced questions (range0-10, (with a score of 0 = None and 10 = Completely) ) how sad are you feeling?in two phases: a. preoperatively, b) in PACU
Evaluating Patients' Sedation | Perioperatively
  Evaluation with Richmond Agitation-Sedation Scale (RASS scale, range +4 to -5, (with a score of -5 = unarousable and +4 = violent, immediate danger for the staff) ).
Evaluating Patients' Sedation | Perioperatively
  Evaluation with Bispectral index (BIS, range 0-100). A BIS score quantifies changes in the electrophysiologic state of the brain during anesthesia. In patients who are awake, a typical BIS score is 90 to 100. Complete suppression of cortical activity results in a BIS score of 0, known as a flat line. Lower numbers indicate a higher hypnotic effect. Overall, a BIS value below 60 is associated with a low probability of response to commands.
Evaluating pain levels between the 2 protocols with scales in PACU | 1 day during hospitalization
  Evaluating perioperative pain levels between the two protocols with scale such as Visual analogu pain scale (VAS, range 0-10, (with a score of 0 = None and 10 = severe pain) ) in PACU
Evaluating stress levels between the 2 protocols with scales | 1 day during hospitalization
  Evaluating perioperative stress levels between the two protocols with scale, such as three self-experienced questions (range0-10, (with a score of 0 = None and 10 = Completely) ) how stressed are you feeling, in two phases: a. preoperatively, b) in PACU
Evaluating stress levels between the 2 protocols with scales | 1 day during hospitalization
  Evaluating perioperative stress levels between the two protocols with scale, such as three self-experienced questions (range0-10, (with a score of 0 = None and 10 = Completely) ) how optimistic are you feeling, in two phases: a. preoperatively, b) in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Konstantinou, RN, PhD, Study Director — National and Kapodistrian University of Athens
Locations (1):
- "Saint Savvas" Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapritsou M, Bozas E, Stavrianos S, Salatas K, Plastiras A, Pistolas K, Fyrfiris N, Kotrotsiou M, Konstantinou EA. The Total Intra Venous Anesthesia Effect Versus Volatile Anesthesia, on Stress and Pain Levels, in Patients Undergoing Breast Reconstruction in Ambulatory Surgery Center Total Intra Venous Anesthesia Protocol and Stress Response. Biol Res Nurs. 2024 Jan;26(1):91-100. doi: 10.1177/10998004231194571. Epub 2023 Aug 9. PMID 37559349